CLINICAL TRIAL: NCT00855140
Title: Acupuncture for the Treatment of Insomnia - A Pilot Study
Brief Title: Acupuncture for the Treatment of Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ronald M. Glick, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21AT004429-01A1 (NIH); R21AT004429 (NIH)
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Primary Insomnia
Keywords: Insomnia; Primary insomnia; Insomnia disorder; Acupuncture
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects were unaware of whether they were receiving verum or sham treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham acupuncture (Placebo Comparator): Sham acupuncture at non-active acupuncture points, using the Park Sham Device
  Interventions: Other: Acupuncture
- Verum Acupuncture (Experimental): Acupuncture following a specific TCM-based protocol
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture, derived from the TCM literature, specific for insomnia

SUMMARY:
Insomnia is a common and disabling condition associated with psychiatric and medical comorbidities and often persists despite currently available treatments. Acupuncture has been reported to benefit individuals with insomnia and can decrease hyperarousal. This blinded RCT will investigate the impact of a standardized acupuncture protocol on insomnia, daytime symptoms, and hyperarousal.

DETAILED DESCRIPTION:
Insomnia is a common problem that is disabling and that frequently persists despite available medical and behavioral approaches. It is associated significant psychiatric and medical comorbidities and high medical and societal costs. Benzodiazepine receptor agonists (BzRA's) and cognitive behavioral therapies are common treatments, but despite these, insomnia remains a pervasive problem. Complementary and alternative medicine (CAM) treatments are being used widely for the treatment of insomnia, but many of these modalities have sparse research support. There are numerous reports in the Traditional Chinese Medicine (TCM)literature of dramatic benefits of acupuncture for the treatment of insomnia, but carefully designed studies are limited. Insomnia has been associated with hyperarousal and acupuncture has documented effects on autonomics with a shift towards parasympathetic predominance. In consultation with experts in acupuncture and TCM, we developed a protocol for the treatment of insomnia and have used it clinically with good success.

We will be conducting a 3-year exploratory pilot randomized-controlled blinded trial (RCT) of this protocol on 56 adults with insomnia disorder, utilizing a control condition involving placement of placebo needles. We seek to determine the effect size of this acupuncture intervention in comparison to the control condition in preparation for a more definitive study, with the future primary aim to determine if acupuncture is effective and well tolerated in the treatment of insomnia. Measures will include self-report and objective measures of sleep quality and duration including polysomnography (PSG). Secondary-exploratory aims will be to determine the impact of this acupuncture protocol on daytime symptoms of insomnia such as fatigue, anxiety, and depression as well as to explore the impact of acupuncture on self-report and objective measures of hyperarousal.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-60;
2. Ability to speak, read, and write English;
3. Insomnia disorder, as defined by RDC, of 3 months or greater duration.

Exclusion Criteria:

1. Presence of serious psychiatric Axis I DSM-IV disorders such as bipolar or psychotic disorders-as individuals with conditions may respond differently than insomnia disorder to the acupuncture intervention, potentially confounding the results;
2. Active suicidal ideation or active psychosis, as this may present a concern regarding safety for a subject's participation in this study;
3. Presence of depressive or anxiety disorders of moderate or greater severity based on either HAM-D scores or HAM-A scores of 14 or greater;
4. Presence of unstable medical conditions commonly associated with significant sleep disturbance, e.g. uncompensated congestive heart failure, as this would not be expected to respond to the acupuncture intervention;
5. Presence of other sleep disorder, such as periodic limb movement disorder or sleep apnea, as these conditions would require other medical treatment-this will be based on known history of sleep disorder or findings on screening PSG of apnea-hypopnea index of > 10 or periodic limb movement index of >10;
6. Alcohol use > 14 beverages/week, as this may impact on response to the intervention and assessment measures;
7. Ongoing use of any recreational drugs;
8. Ongoing use of benzodiazepines, prescription hypnotic medication, over-the-counter hypnotic medication, or nutritional supplements with purported hypnotic effects;
9. Ongoing use of other psychotropic medication, such as psychostimulants, or antipsychotics;
10. Caffeine use > the equivalent of 5 cups of coffee/day;
11. Pregnancy, as the safe use of acupuncture in pregnancy has not been established;
12. Active malignancy, autoimmune condition, or treatment with immunosuppressive drugs;
13. Presence of coagulopathy or use of anticoagulant medication;
14. Active involvement in any psychotherapy or other treatment specifically directed towards insomnia;
15. Prior experience with acupuncture treatment in the last 6 months or prior participation in an acupuncture research study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency on polysomnography | Baseline and post-intervention
  PSG is the "gold standard" objective measure of sleep, which complements in-home diary measures and actigraphy. PSG provides objective physiologic data under controlled, albeit artificial (laboratory) conditions and is considered an essential component of demonstrating the efficacy of both drug and non-pharmacologic treatments of insomnia.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, EOI, & 3 months post-tx
  A 19-item questionnaire developed by Buysse et. al. that rates the subject's habitual sleep over the past month(109). The 19 questions are combined into seven clinically-derived component scores, each weighted equally from 0-3. The seven component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality.
Insomnia Severity Index (ISI) | Baseline, EOI, & 3 months post-tx
  A 7-item survey which rates satisfaction with different aspects of sleep over the prior two weeks on a 0-4 Likert scale for a total score of 28, with a higher score reflecting greater severity of insomnia(126). Criteria are specified to categorize response into one of four severity groups, with a change of one level considered significant.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | Baseline, EOI, & 3 months post-tx
  evaluates the tendency to fall asleep during various daytime activities
Multidimensional Fatigue Inventory (MFI) | Baseline, EOI, & 3 months post-tx
  20-item self-report instrument designed to measure fatigue. It includes 5 subscales addressing dimensions of General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation, and Reduced Activity.
Inventory for Depressive Symptomatology-Self-Rated (IDS-SR) | Baseline, EOI, & 3 months post-tx
  28-item self-rating scale for depressive symptoms with each item rated on a 0-3 Likert scale with higher scores representing increasing depressive symptoms
State version of the Spielberger State-Trait Anxiety Inventory (STAI-s) | Baseline, EOI, & 3 months post-tx
  validated measure of state anxiety in which subjects are asked to rate the severity of mood and anxiety symptoms at this moment, with 20 symptoms rated on a 1-4 Likert scale
The Pre-Sleep Arousal Scale (PSAS) | Baseline, EOI, & 3 months post-tx
  16-item self-report questionnaire with two 8-question subscales representing the cognitive and somatic components of arousal
Pittsburgh Sleep Diary (PghSD) and actigraphy recording | Baseline, EOI, & 3 months post-tx
  A daily record of sleep quality and sleep-related behaviors that includes bedtime and waketime portions.
Autonomic arousal as measured by HRV & Q-EEG during sleep recording | Baseline & EOI
  A standardized battery of mild psychological stressors that have been used successfully here at the University of Pittsburgh in studies of autonomic reactivity and which we are currently using to study the effects of CAM interventions on autonomic reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Glick, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Center for Integrative Medicine at UPMC Shadyside, Pittsburgh, Pennsylvania, United States